CLINICAL TRIAL: NCT07097220
Title: Effects of Different Anesthetic Techniques on Intraoperative and Postoperative Pain Levels and Cognitive Function in Patients Undergoing Hepatectomy for Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital, Qingchun Campus, Zhejiang University School of Medicine, (Other Government)
Responsible Party: Principal Investigator, Juhui Chen, Principal Investigator, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: No. 2025-0355
Record Dates: First submitted 2025-06-30; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Liver Cancer; Hepatectomy; Anesthesia Techniques; Postoperative Pain; Cognitive Dysfunction; Epidural-general Anesthesia
MeSH Terms: conditions — Liver Neoplasms; Pain, Postoperative; Cognitive Dysfunction | interventions — Anesthesia, General; Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia group (Experimental): In the General Anesthesia (GA) group (n = 59), patients received combined intravenous-inhalation general anesthesia. Anesthesia induction was performed using propofol and remifentanil, followed by maintenance with sevoflurane to ensure adequate anesthetic depth and hemodynamic stability throughout the procedure.
  Interventions: Drug: General Anesthesia (GA) group
- General-Epidural Anesthesia group (Experimental): In the General-Epidural Anesthesia (GEA) group (n = 47), patients received the same general anesthesia protocol as the GA group, in addition to epidural anesthesia. An epidural catheter was placed preoperatively at the T7-T9 vertebral level using a midline approach under strict aseptic conditions. Following successful catheterization and confirmation of proper placement, a continuous intraoperative infusion of 0.25% ropivacaine was administered via the epidural route to provide segmental analgesia and reduce intraoperative opioid requirements.
  Interventions: Drug: General-Epidural Anesthesia (GEA) group

INTERVENTIONS:
Drug: General Anesthesia (GA) group — In the General Anesthesia (GA) group (n = 59), patients received combined intravenous-inhalation general anesthesia. Anesthesia induction was performed using propofol and remifentanil, followed by maintenance with sevoflurane to ensure adequate anesthetic depth and hemodynamic stability throughout the procedure.
  Arms: general anesthesia group
Drug: General-Epidural Anesthesia (GEA) group — In the General-Epidural Anesthesia (GEA) group (n = 47), patients received the same general anesthesia protocol as the GA group, in addition to epidural anesthesia. An epidural catheter was placed preoperatively at the T7-T9 vertebral level using a midline approach under strict aseptic conditions. Following successful catheterization and confirmation of proper placement, a continuous intraoperative infusion of 0.25% ropivacaine was administered via the epidural route to provide segmental analgesia and reduce intraoperative opioid requirements.
  Arms: General-Epidural Anesthesia group

SUMMARY:
To evaluate the effects of general anesthesia (GA) versus combined general and epidural anesthesia (GEA) on postoperative pain, cognitive dysfunction (POCD), hospital stay, and recovery quality in liver cancer patients undergoing hepatectomy.

A retrospective analysis of 80 liver cancer patients was conducted, categorized by analgesic adequacy, pain recovery, and POCD incidence: adequate vs. inadequate analgesia (n=50 vs. n=30), favorable vs. delayed pain recovery (n=36 vs. n=44), and POCD vs. non-POCD (n=42 vs. n=38). Based on these results, a prospective study (April 2024-April 2025) enrolled patients scheduled for elective hepatectomy, assigned to the GA group (n=59) or GEA group (n=47). Primary outcomes included intraoperative analgesic consumption, postoperative VAS pain scores, MoCA cognitive scores, hospital stay length, and adverse event rates.

DETAILED DESCRIPTION:
Compared to GA alone, combined epidural-general anesthesia provides better perioperative pain control, reduces POCD risk, shortens hospitalization, and enhances recovery. GEA is a preferable anesthetic approach for liver cancer surgery.

ELIGIBILITY:
* Inclusion Criteria:
* Histologically or radiologically confirmed primary liver cancer (HCC or cholangiocarcinoma)
* Scheduled for elective open or laparoscopic radical hepatectomy
* Age 18-75 years
* ASA Physical Status I-III
* Child-Pugh class A or B liver function
* Normal preoperative MoCA score (≥26)
* Willing to participate and provide informed consent
* Exclusion Criteria:
* Severe cardiovascular, pulmonary or renal disease (ASA IV/V)
* Chronic pain disorders or preoperative opioid use (>3 months)
* Known neurologic/psychiatric conditions (dementia, stroke, epilepsy)
* Concurrent major procedures (e.g., vascular resection)
* Intraoperative conversion to palliative surgery
* Massive intraoperative hemorrhage (>2000 mL)
* Coagulopathy (INR >1.5 or platelets <50×10⁹/L)
* Spinal abnormalities precluding epidural catheterization
* Pregnancy or lactation
* Allergy to local anesthetics or study medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Cognitive Dysfunction (POCD) | Baseline (preoperative), POD1 (24±4h), POD3 (72±6h)
  Percentage of patients with:
  MoCA score <26 at postoperative assessment OR
  ≥2-point decrease from preoperative baseline (Assessed using Montreal Cognitive Assessment, 30-point scale)
Postoperative Pain Intensity | 2h, 6h, 12h, 24h, 48h postoperatively
  Mean pain scores measured by:
  Visual Analog Scale (VAS)
  10cm scale (0=no pain, 10=worst pain)

SECONDARY OUTCOMES:
Intraoperative Opioid Consumption | Anesthesia induction to extubation
  Total remifentanil dose administered:
  Measured in micrograms (μg)
  Recorded from anesthesia machine
Hospital Length of Stay | Up to 30 days post-surgery
  Duration from surgery end to discharge:
  Measured in days
  From electronic medical records
Adverse Event Incidence | 0-72 hours postoperatively
  Percentage of patients with:
  Nausea/vomiting
  Delirium (CAM-positive)
  Other complications

OTHER OUTCOMES:
Intraoperative Analgesic Adequacy | Entire surgical duration
  Percentage of patients with:
  Grade I (adequate) vs
  Grades II-IV (inadequate) analgesia (Per Supplementary Table S1 criteria)
Surgical Stress Correlation | Intraoperative period
  Pearson correlation coefficients between:
  Anesthesia technique (GA/GEA)
  Blood loss (mL)
  Surgery duration (min)

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China